CLINICAL TRIAL: NCT02840565
Title: A Double-blind, Randomised, Placebo-controlled Study to Evaluate the Tolerability, Pharmacokinetics and Pharmacodynamics of Six Multiple Rising Dose Regimens of BIA 5-453 in Healthy Male Volunteers
Brief Title: Tolerability, Pharmacokinetics and Pharmacodynamics of Six Multiple Rising Dose Regimens of BIA 5-453
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-5453-102; 2007-004142-33 (EudraCT Number)
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Hypertension; Chronic Heart Failure
MeSH Terms: conditions — Hypertension | interventions — etamicastat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- BIA 5-453 25 mg or placebo (Experimental): Multiple oral doses of BIA 5-453 25 mg or placebo were administered once daily for 10 days to subjects in fasting conditions.
  Interventions: Drug: BIA 5-453; Drug: Placebo
- BIA 5-453 50 mg or placebo (Experimental): Multiple oral doses of BIA 5-453 50 mg or placebo were administered once daily for 10 days to subjects in fasting conditions.
  Interventions: Drug: BIA 5-453; Drug: Placebo
- BIA 5-453 100 mg or placebo (Experimental): Multiple oral doses of BIA 5-453 100 mg or placebo were administered once daily for 10 days to subjects in fasting conditions.
  Interventions: Drug: BIA 5-453; Drug: Placebo
- BIA 5-453 200 mg or placebo (Experimental): Multiple oral doses of BIA 5-453 200 mg or placebo were administered once daily for 10 days to subjects in fasting conditions.
  Interventions: Drug: BIA 5-453; Drug: Placebo
- BIA 5-453 400 mg or placebo (Experimental): Multiple oral doses of BIA 5-453 400 mg or placebo were administered once daily for 10 days to subjects in fasting conditions.
  Interventions: Drug: BIA 5-453; Drug: Placebo
- BIA 5-453 600 mg or placebo (Experimental): Multiple oral doses of BIA 5-453 600 mg or placebo were administered once daily for 10 days to subjects in fasting conditions.
  Interventions: Drug: BIA 5-453; Drug: Placebo

INTERVENTIONS:
Drug: BIA 5-453 — Presented as blue hard gelatine capsules (size 2) of 1 mg, 10 mg and 50 mg for oral administration
  Other Names: Etamicastat
Drug: Placebo — The composition of the placebo is qualitatively the same but without BIA 5-453 pharmaceutical active ingredient.

SUMMARY:
The purpose of this study is to assess the tolerability of BIA 5-453 after six multiple rising dose regimens of BIA 5-453.

DETAILED DESCRIPTION:
Two centres, double-blind, randomised, placebo-controlled study of six dosage regimens of BIA 5-453 in six groups of healthy male subjects.

In each group, the study consisted of a 10-day multiple-dose period. Progression to the next dose level only occurred if the previous dose level was considered to be safe and well tolerated. An appropriate interval separated the investigation of doses to permit a timely review and evaluation of safety data (including plasma exploratory pharmacokinetics) prior to proceeding to a higher dose level.

ELIGIBILITY:
Inclusion Criteria:

1. A signed and dated informed consent form before any study-specific screening procedure was performed.
2. Aged between 18 and 45 years, inclusive.
3. Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs and digital 12-lead ECG.
4. Nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history. Must have been able to abstain from smoking during the inpatient stay.
5. Have a high probability for compliance with and completion of the study.

Exclusion Criteria:

Medical History

1. Any significant cardiovascular (e.g. hypertension), hepatic, renal, respiratory (e.g. childhood asthma), gastrointestinal, endocrine (e.g. diabetes, dyslipidemia), immunologic, dermatological, haematological, neurologic, or psychiatric disease.
2. Acute disease state (e.g., nausea, vomiting, fever, diarrhoea) within 7 days before study Day1.
3. History of drug abuse within 1 year before study Day1.
4. History of alcoholism within 1 year before Day1. Consumption of more than 50 g of ethanol per day (12.5 cL glass of 10° [10%] wine = 12 g; 4 cL of aperitif, 42° [42%] whiskey = 17 g; 25 cL glass of 3° [3%] beer = 7.5 g; 25 cL glass of 6° [6%] beer = 15 g
5. History of any clinically important drug allergy.

   Physical and Laboratory Findings
6. An automatic ECG QTc interval reading at screening or enrolment >450 ms.
7. Positive serologic findings for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibodies.
8. Positive findings of urine drug screen (eg, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, MDMA [3,4-methylenedioxy-methamphetamine; ecstasy]).

   Prohibited treatments
9. Prohibited Treatments: use of any investigational drug within 90 days or prescription drug within 30 days before investigational medical product (IMP) administration.
10. Consumption of any caffeine-containing products (e.g., coffee, tea, chocolate, or soda) in excess of 6 cups per day (or equivalent), of grapefruit, grapefruit-containing products, or alcoholic beverages within 72 before study day -1.
11. Use of any over-the-counter drugs including herbal supplements (except for the occasional use of acetaminophen [paracetamol], aspirin and vitamins ≤100% recommended daily allowance) within 7 days before IMP administration.
12. Donation of blood (ie 450 ml) within 90 days before study Day1.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2007-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Percent of subjects with at least one adverse event | through study completion, an average of 10 days
Percent of subjects by dose group with at least one treatment-emergent adverse event (TEAEs) | through study completion, an average of 10 days
  Treatment-emergent adverse events are adverse events that occurred either in the 72 hours after dosing or that was present prior to dosing but exacerbated within 72 hours after dosing.

IPD SHARING:
Plan to Share IPD: Undecided